CLINICAL TRIAL: NCT04893681
Title: Proof-of-concept Randomized Controlled Trial to Evaluate Dental Caries Preventive Effects of Fluoridated Bottled Water
Brief Title: Water From Bottles to Establish Strong Teeth
Acronym: waterBEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Tulane University (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-3273; UG3DE029169 (NIH); 21-017-E (Other: NIDCR study protocol number)
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries in Children
Keywords: Fluorides

STUDY DESIGN:
Intervention Model Description: Block randomized, double-masked, placebo controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be managed by the a Data Management System which will execute three tasks:
  1. Study participants' treatment group allocation will be stored in a dataset accessible only to the masked data manager
  2. A separate dataset will record unique identification codes that will be affixed as labels to 5-gallon bottles of water; the same dataset will also record the public water supply used to fill the bottle (New Bern or North Lenoir). After the barcode label is affixed, the processing slip indicating the bottle's source of water (New Bern or North Lenoir), will be removed, thereby masking the contents.
  3. When new water bottles are to be delivered to a study participant's dwelling, the Data Management System will execute a bottle allocation routine that will retrieve the study participant's study group assignment and select from the supply of masked bottles the necessary number of masked bottles that conform with the study participant's treatment group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoridated bottle water (Experimental): 5-gallon bottles containing water from the New Bern Water Resources Division's Black Creek aquifer which contains naturally-occurring fluoride in a concentration of approximately 0.8 mg/L F
  Interventions: Other: Fluoridated bottled drinking water
- Non-fluoridated bottled water (Placebo Comparator): 5-gallon bottles containing water from the North Lenoir Water Corporation's Black Creek aquifer which contains a negligible concentration of fluoride.
  Interventions: Other: Non-fluoridated drinking water

INTERVENTIONS:
Other: Fluoridated bottled drinking water — Study participants are asked to consume study water, as frequently and in amounts as necessary or desired, whenever they drink water (e.g., as plain water or mixed with other ingredients) or use water in food preparation.
  Arms: Fluoridated bottle water
Other: Non-fluoridated drinking water — Study participants are asked to consume study water, as frequently and in amounts as necessary or desired, whenever they drink water (e.g., as plain water or mixed with other ingredients) or use water in food preparation.
  Arms: Non-fluoridated bottled water

SUMMARY:
The waterBEST study is a proof-of-concept, randomized, double-masked, placebo controlled, parallel group study evaluating dental caries-preventive effects of fluoridated bottled water compared to non-fluoridated bottled water in 4-year-old children.

DETAILED DESCRIPTION:
This is a proof-of-concept, randomized, double-masked, placebo controlled, parallel group study evaluating dental caries-preventive effects of fluoridated bottled water compared to non-fluoridated bottled water in 4-year-old children. Children will be allocated at random to receive either fluoridated or non-fluoridated sourced from two local public water systems. The water will be packaged into 5-gallon bottles and delivered to households during a 3½ year intervention period. During the intervention period, parents/guardians/caregivers will be interviewed quarterly to monitor children's general health and a dental screening will be conducted annually. Children's fingernail and toenail clippings will be collected annually and analyzed to determine the fluoride content as a biomarker of total fluoride intake. Dental caries experience, the primary endpoint, will be determined once in a dental examination conducted by a study dentist close to the time of the child's 4th birthday. For the primary aim, a least-squares, generalized linear model will estimate efficacy and its one-tailed, upper 80% confidence limit using the number of decayed, missing and filled primary tooth surfaces as the dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* The parent/guardian/caregiver understands and consents to procedures described in parental permission and consent form.
* Child is aged 2 months to 6 months at the screening visit.
* Child either drinks water (either plain water, or water mixed with something) or is expected to drink water by their first birthday, as reported by the parent/guardian/caregiver at the screening visit.

Exclusion Criteria:

* The child's primary dwelling at the screening visit has tap water that contains >0.60 mg/L F and the parent/guardian/caregiver expresses a preference that the child drink tap water, not bottled water, for the child's first four years of life. For children who live at more than one dwelling, the primary dwelling is defined as the one at which they usually sleep at least four nights per week.
* Child has serious illness/es requiring frequent inpatient hospitalization, as reported by the parent/ guardian/caregiver at the screening visit.
* Child's birth weight was less than 1,500 g (3 pounds 5 ounces).
* Child's gestational age was less than 34 weeks.
* Child uses fluoride supplements, as reported by the parent/ guardian/caregiver at the screening visit.
* Parent/guardian/caregiver states at the screening visit the child will initiate fluoride supplementation before the child's 4th birthday
* The parent/ guardian/caregiver anticipates that the child will move to an address more than 30 miles from Kinston, NC before the child's 4th birthday.
* The investigators determine that a child living at the same primary dwelling has already been enrolled in the study. (This means that if two or more children fulfilling the inclusion criteria live at the primary dwelling, the parent will be asked to select one such child to be the study participant.)
* Anything that, in the opinion of the principal investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
dmfs index | Dental examination in year 4
  The number of primary tooth surfaces that are decayed, missing or filled will be enumerated during dental examinations of children near the time of their 4th birthday. Decay will be assessed clinically at the threshold of macroscopic enamel loss, as per criteria defined by the International Caries Detection and Assessment System. Five surfaces per tooth will be enumerated in all primary teeth (maximum = 20 teeth per child), yielding a count of affected surfaces that can range from 0 (no dental caries experience) to 100 (worst possible extent of dental caries experience). The lower-case abbreviation "dmfs" signifies disease in the primary dentition, a convention used to distinguish it from equivalent measures for the permanent dentition, where an uppercase abbreviation is used, as defined for the National Library of Medicine's Medical Subject Heading heading "DMF Index".

SECONDARY OUTCOMES:
Fluoride content of fingernail and toenail biospecimens | Up to three years after randomization.
  Fluoride content of fingernail and toenail clippings will provide a biomarker of total fluoride intake at intervals of 1, 2 and 3 years after randomization. Fluoride content will be measured in mg/kg using a hexamethyldisiloxane-facilitated diffusion assay of nail clippings collected from study subjects.
Adverse events | Through study completion, an average of 42 months.
  Number of adverse events, sub-classified according to whether or not the event is serious, and whether or not the event is related (either possibly, probably or definitely) to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slade, BDSc, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Division of Pediatric and Public Health, UNC Adams School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Derived] Sanders AE, Divaris K, Godebo TR, Slade GD. Effect of bottled fluoridated water to prevent dental caries in primary teeth: study protocol for a phase 2 parallel-group 3.5-year randomized controlled clinical trial (waterBEST). Trials. 2024 Mar 5;25(1):167. doi: 10.1186/s13063-024-08000-4. PMID 38443989